CLINICAL TRIAL: NCT01804439
Title: Cardiovascular Risk Factors in the Initial Presentation of Specific Cardiovascular Disease Syndromes: a CALIBER Proposal Using Linked GPRD-MINAP-HES Data
Brief Title: Risk Factors in the Initial Presentation of Specific Cardiovascular Disease Syndromes
Status: Completed | Type: Observational
Sponsor: University College, London (Other)
Responsible Party: Principal Investigator, Harry Hemingway, Professor Harry Hemingway, University College, London
Other Study IDs: CALIBER 12_153R
Record Dates: First submitted 2013-01-08; First posted 2013-03-05 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Heart Diseases; Cardiovascular Diseases; Acute Myocardial Infarction; Unstable Angina; Chronic Stable Angina; Ischemic Stroke; Cerebrovascular Accident; Subarachnoid Hemorrhage; Transient Ischemic Attack; Abdominal Aortic Aneurysm; Peripheral Arterial Disease; Sudden Coronary Death; Ventricular Arrhythmia; Sudden Death; Cardiac Arrest; Heart Failure
Keywords: Heart diseases; Cardiovascular diseases; Coronary heart disease not otherwise specified; Cerebrovascular disorders; Brain diseases; Central nervous system diseases; Nervous system diseases; Atherosclerosis; Arteriosclerosis; Pathologic processes; Acute myocardial infarction; Myocardial infarction; Myocardial ischemia; Infarction; Necrosis; Unstable angina; Chronic stable angina; Stable angina; Angina pectoris; Chest pain; Pain; Signs and symptoms; Ischemia; Ischemic stroke; Hemorrhagic stroke; Stroke; Subarachnoid hemorrhage; Transient ischemic attack; Abdominal aortic aneurysm; Aneurysm; Aortic aneurysm; Aortic aneurysm, abdominal; Aortic diseases; Peripheral arterial diseases; Peripheral vascular diseases; Vascular diseases; Peripheral occlusive diseases; Sudden coronary death; Ventricular arrhythmia; Sudden cardiac death; Cardiac arrest; Heart failure
MeSH Terms: conditions — Heart Diseases; Cardiovascular Diseases; Angina, Unstable; Angina, Stable; Ischemic Stroke; Stroke; Subarachnoid Hemorrhage; Ischemic Attack, Transient; Aortic Aneurysm, Abdominal; Peripheral Arterial Disease; Death, Sudden; Heart Arrest; Heart Failure; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Atherosclerosis; Arteriosclerosis; Pathologic Processes; Myocardial Infarction; Myocardial Ischemia; Infarction; Necrosis; Angina Pectoris; Chest Pain; Pain; Signs and Symptoms; Ischemia; Hemorrhagic Stroke; Aneurysm; Aortic Aneurysm; Aortic Diseases; Peripheral Vascular Diseases; Vascular Diseases; Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CALIBER Healthy Cohort: We will report findings from the CALIBER (CArdiovascular disease research using Linked BEspoke studies and Electronic Records) collaboration where we linked primary care data (from the General Practice Research Database [GPRD]) to three further sources of electronic health records: the Myocardial Ischemia National Audit Project registry (MINAP),cause specific discharge data from Hospital Episodes Statistics (HES) and cause specific mortality from the Office for National Statistics (ONS).

SUMMARY:
Cardiovascular disease (CVD) is an important public health problem that affects millions of people worldwide. Associations between risk factors, such as smoking, dyslipidaemia or hypertension, and prevalent CVD are well documented. However, few studies have investigated associations with onset of disease. The initial manifestation of CVD, for example an episode of unstable angina, is important because it influences the prognosis, the quality of life and the management of disease. Furthermore, the extent to which social deprivation, alcohol consumption or atrial fibrillation affects presentation of CVD is poorly understood and deserves further consideration.

Most previous studies have considered CVD as a single entity. However, differences in aetiology between coronary phenotypes suggest that risk factors may not be shared across specific coronary phenotypes and their relative importance is likely to differ for each phenotype. Gaining knowledge of these differences could provide insights into the pathophysiology of specific forms of CVD and could eventually lead to modification of recommendations for patient management and disease prevention.

We propose to use the linkage of the national registry of coronary events to general practice records in the Clinical Practice Research Database (CPRD), to investigate whether demographic, behavioral, and clinico-metabolic risk factors differentially influence the onset of specific types of CVD.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥30yrs old
* Registered in CPRD practices in England consenting to data linkage
* ≥1 year of up-to-standard pre-study follow-up

Exclusion Criteria:

* History of any of the CVD endpoints considered before study follow-up initiation.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will include all patients aged ≥30yrs old, registered in CPRD practices in England consenting to data linkage, with at least 1 year of up-to-standard pre-study follow-up and no history of any of the CVD endpoints considered. Follow-up for endpoints will commence on the earliest date on which a patient fulfils the criteria, within the period between 1st January 1997 and 25th March 2010.
Sampling Method: Non-Probability Sample
Enrollment: 2240000 (Actual)
Dates: Start 1997-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
First presentation of cardiovascular disease, as specified in description | Study follow-up will commence on the earliest date on which a patient fulfils the criteria for study inclusion within the period between 1st January 1997 and 25th March 2010 (maximum of 13 years after enrolment).
  First occurrence of the following fatal or non-fatal cardiovascular outcomes: acute myocardial infarction, unstable angina, stable angina, ischemic stroke, hemorrhagic stroke, subarachnoid hemorrhage, transient ischemic attack, abdominal aortic aneurysm, peripheral arterial disease, sudden cardiac death, heart failure

SECONDARY OUTCOMES:
Non CVD specific deaths | Same as for primary outcomes (maximum of 13 years after follow-up start)
  Death from non CVD, that is, excluding deaths related to the primary endpoints.

OTHER OUTCOMES:
Cardiovascular heart disease and fatal cardiovascular disease | Same as for primary endpoint (maximum of 13 years after follow-up start)
  Cardiovascular heart disease: combination of MI and unheralded coronary death. Cardiovascular disease: combination of fatal cardiovascular heart disease and stroke of any type.
  Fatal cardiovascular disease: combination of fatal coronary heart disease and fatal cardiovascular death.

REFERENCES:
- [Derived] Dinesh Shah A, Langenberg C, Rapsomaniki E, Denaxas S, Pujades-Rodriguez M, Gale CP, Deanfield J, Smeeth L, Timmis A, Hemingway H. Type 2 diabetes and incidence of a wide range of cardiovascular diseases: a cohort study in 1.9 million people. Lancet. 2015 Feb 26;385 Suppl 1:S86. doi: 10.1016/S0140-6736(15)60401-9. PMID 26312908
- [Derived] Shah AD, Langenberg C, Rapsomaniki E, Denaxas S, Pujades-Rodriguez M, Gale CP, Deanfield J, Smeeth L, Timmis A, Hemingway H. Type 2 diabetes and incidence of cardiovascular diseases: a cohort study in 1.9 million people. Lancet Diabetes Endocrinol. 2015 Feb;3(2):105-13. doi: 10.1016/S2213-8587(14)70219-0. Epub 2014 Nov 11. PMID 25466521